CLINICAL TRIAL: NCT02572973
Title: Acoustic Neuromodulation (ANM) for Youth With Anxiety Disorders: A Pilot Study
Brief Title: Acoustic Neuromodulation (ANM) for Youth With Anxiety Disorders
Acronym: ANM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Rate of recruitment deemed insufficient by study sponsor
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: The Hartwell Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1403014928
Record Dates: First submitted 2015-06-24; First posted 2015-10-09 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Separation Anxiety Disorder; Generalized Anxiety Disorder; Social Phobia
MeSH Terms: conditions — Anxiety, Separation; Generalized Anxiety Disorder; Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Treatment (Active Comparator): The Acoustic Neuromodulation (ANM) active treatment intervention is a non-invasive form of therapy in which certain sounds at certain intervals are delivered to a subject through headphones five times over the course of two weeks. The sounds are delivered for 12 minutes at each session. The level of sound during Sound Stimuli (SS) presentation is relatively low (20-40 decibels), and the volume level can be adjusted downward if the subject requests it. The active intervention sounds used in the trial couple sequential frequencies to the base frequency in a nonlinear (exponential) manner following a special algorithm developed by Dr. Izvarina. This algorithm varies both the rate of change and duration of the overlaying modulation that is presented to the brain.
  Interventions: Other: Acoustic Neuromodulation (ANM)
- Non-Active Placebo (Placebo Comparator): The Acoustic Neuromodulation (ANM) treatment intervention is a non-invasive form of therapy in which certain sounds at certain intervals are delivered to a subject through headphones five times over the course of two weeks. The sounds are delivered for 12 minutes at each session. The placebo sounds used in this trial mimic the active sounds, but instead of using nonlinear modulation, they are coupled to the base frequency in a linear manner. Both the sequence used as well as the rate of change and duration of this overlaying modulation are the same as that used for the active sounds. The only difference is use of a linear algorithm for the placebo sounds and a nonlinear (exponential) algorithm for the active sounds.
  Interventions: Other: Acoustic Neuromodulation (ANM)

INTERVENTIONS:
Other: Acoustic Neuromodulation (ANM) — The purpose of this study is test the safety of the Acoustic Neuromodulation (ANM) treatment and see what effects it has on your child's anxiety symptoms. Observation and anecdotal evidence suggest that this is an effective intervention for anxiety disorders. This is the first research study to test this theory, and could lead to more robust studies in the future. This study intends to assess the efficacy of this type of intervention for children with an anxiety disorder. As this is only a pilot study, the results will also inform the design and execution of future research on this treatment. We hope to add to the growing literature supporting novel treatment approaches for affected individuals.

SUMMARY:
The acoustic neuromodulation trial (ANM-T) is a two-phase, single-site, pilot randomized clinical trial examining the feasibility of completing a larger scale efficacy study of a novel treatment of non-linear modulated acoustic stimuli to reduce anxiety severity in youth with anxiety disorders. The primary objective is to establish the feasibility of a blinded randomized controlled trial of ANM for childhood anxiety disorders.

DETAILED DESCRIPTION:
The acoustic neuromodulation trial (ANM-T) is a two-phase, single-site, pilot randomized clinical trial examining the feasibility of completing a larger scale efficacy study of a novel treatment of non-linear modulated acoustic stimuli to reduce anxiety severity in youth with anxiety disorders. Phase I involves a randomized controlled trial comparing active acoustic neuromodulation to a non-active acoustic stimuli (Placebo or PBO) in youth ages 7-17 years with at least one of the following primary DSM-5 diagnoses: separation anxiety disorder (SAD), social anxiety disorder and generalized anxiety disorder (GAD).

Additionally, this study will include up to ten healthy volunteer participants in order for study staff to be appropriately trained to administer the EEG. Furthermore, three pilot cases will be completed at the start of data collection to ensure effective delivery of all study procedures and maintenance of blind during the acute study phase. Phase II is a 3-month treatment maintenance period for Phase I responders. Phase I non-responders to PBO will be offered active open treatment. Assessments will include those that will likely be used in a larger efficacy trial including parent on child report, and child self report, and blinded independent evaluator ratings of the primary outcomes. In addition, in an effort to assess over all feasibility, monthly recruitment rate, number of consents signed, subjects randomized, rate of adherence to the treatment protocol, safety of the intervention and control conditions, patient and family acceptability of the treatment and assessment protocols will be evaluated. Study Phases Entry Gates: 30 subjects ages 7-17 years will be enrolled, using a multiple gating procedure designed to ensure that subjects enrolled evidence a stable, pervasive anxiety diagnosis at the start of treatment.

* Gate A is a 20-minute semi-scripted telephone screening procedure to elicit preliminary inclusion/exclusion information and to provide additional information to the caller.
* Gate B is a screening assessment that determines "caseness".

After completing informed consent participants and their parents will complete standard questionnaires and will be interviewed to establish that the child meets all inclusion and no exclusion criteria and are medically safe to complete the study (clearance from the pediatrician and pregnancy test for menstruating females). This visit will be videotaped and will last approximately 2.5 hours.

-Gate C is a baseline assessment of anxiety severity and randomization visit and takes approximately 2.5 hours and will be videotaped. All subjects will be recruited and screened and enrolled by investigators at the Weill Cornell Medical College.

Phase I: Phase I is a 6-week randomized (1:1) controlled comparison of ANM and PBO. Subjects will come in for 20-minute treatment sessions approximately every other day for 2 weeks (5 days in 2 weeks). At each study treatment visit the study coordinator will collect a brief interim history of anxiety symptoms and adverse events prior to treatment. Formal outcome assessment by the blind independent evaluator (IE) will be collected at week 6.

Phase II: Phase II is a 17 week treatment maintenance phase (from week 7 to 24). At this stage, ALL PARTICIPANTS will begin active treatment. Active responders from phase 1 will be monitored for the durability of the treatment response. Non-responders to the active treatments will be given a second chance to elicit a response. Non-responders to control treatment will have a full course of the active treatment. Control treatment responders will be given the chance to respond to active treatment. At each study visit the coordinator will collect an interim history and adverse events. Formal outcome assessment by a blind independent evaluator will occur at weeks 12 and 24

ELIGIBILITY:
Inclusion Criteria:

* Ages 7-17 years inclusively (i.e., must be at least 7 years) at the point of consent
* Primary DSM 5 diagnosis of SepAD, SocAD, or GAD on the ADIS-RLV (Gate B).
* Anxiety severity of moderate or greater (CGI-S >3 and functional impairment (CGAS score of <60) (Gate C).

Exclusion Criteria:

* Estimated child Full Scale IQ < 80, as measured by the vocabulary and block design subtests of the WISC-III) (Gate B). If a potential subject has a verified IQ score in the three years prior to enrollment as measured by the WISC-III, IIIR, K-ABC, or Stanford-Binet no IQ assessment is required.
* Child meets criteria for current primary or co-primary Panic Disorder, OCD, PTSD, conduct disorder or substance abuse (Gate B).
* Child meets criteria for Major Depressive Disorder at greater severity than anxiety disorder (Gate B). d. Subjects with the following lifetime psychiatric disorders will be excluded: bipolar disorder, PDD (Asperger's, autism), MDD with psychosis, schizophrenia, and schizoaffective disorder (Gate B).
* Current use of psychotropic medication or clinical indication for use of psychotropic medication (except for youth entering on a stable psychostimulant regimen for ADHD) (Gates A, B).
* Recent treatment with psychotropic medication within 6 weeks of study entry for fluoxetine, within 2 weeks for other SSRIs, and within 4 weeks for neuroleptics (Gates A, B).
* Child has failed an adequate trial of CBT for anxiety within the previous 2 years (at least 10 treatment sessions over a period of less than 1 year conducted by a licensed provider of CBT) (Gates A, B).
* Child has a major neurological disorder, a major medical illness or hearing impairment that requires a prohibited episodic or chronic systemic medication or that would interfere with participation in the study (e.g., frequent hospitalizations, frequent school absences) (Gates A, B).
* Child is pregnant as indicated by history or a positive pregnancy test at Gate B. Sexually active girls must agree to use an effective form of birth control, either hormonal (BCP, Depo-Provera or Norplant), spermicide (foam or vaginal suppository) or a barrier method (condoms, diaphragm, cervical cap) or a combination of barrier/spermicide contraception in order to participate in the study.
* Child poses a significant risk for dangerousness to self or to others (Gates A, B, C).
* Child or parent is non-English speaking (unable to complete measures, IE ratings or treatment without the assistance of a translator) (Gates A, B). NYSPI and UCLA may recruit Spanish speaking subjects.
* Child is a victim of ongoing or previously undisclosed child abuse requiring new department of social service report or ongoing department of social service supervision (Gate B).
* Child, for any reason, has missed more than 50% of school days in the 2 months preceding randomization. Home schooling does not require exclusion from the study under this exclusion criterion. Ambiguous cases are referred to Caseness Panel to avoid truncating the severity range differently across sites (Gates A, B).
* Child has a history of seizures

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Anxiety Disorders Interview Schedule (ADIS) | 12 weeks. The ADIS will be measured at Wk 0, Wk 6, and Wk 12.
  The ADIS will be measured to to establish the efficacy of ANM to placebo in reducing anxiety symptoms and associated disability.

SECONDARY OUTCOMES:
Electroencephalogram (EEG) | 12 Weeks. EEGs will be administered at Wk 0, Wk 1, Wk 2, Wk 4, Wk 6, Wk 7, Wk 8, Wk 10 and and Wk 12.
  The EEG uses original software to calculate spectral density of bioelectrical brain activity in different frequency ranges, and power of heart pulse spectrum in low frequency and high frequency ranges, in order to characterize the vagal-sympathetic balance of a given subject. The EEG is administered to monitor changes over course of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Walkup, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No